CLINICAL TRIAL: NCT07159477
Title: TEN TENE TEMASIN BABA-BEBEK BAĞLANMASINA ETKİSİ: RANDOMİZE KONTROLLÜ ÇALIŞMA
Brief Title: Effect of Skin-to-Skin Contact on Father-Infant Bonding: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Çanakkale Onsekiz Mart University (Other)
Responsible Party: Principal Investigator, Nazli Emel Ozer Yurdal, Principal Investigator, Çanakkale Onsekiz Mart University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2023-YÖNP-0008
Record Dates: First submitted 2025-08-15; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Newborn Basic Care Training; Newborn Infant; Attachment; Bonding
Keywords: Bonding, Fathers, Newborn.

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fathers who received standard care (SC): (No Intervention): No intervention was given to the fathers in this group according to their order of participation in the study. In the second interview with these fathers, after the data were collected, they were given information and brochures about skin-to-skin contact.
- Early skin-to-skin contact group (ESSC): (Experimental): Fathers in this group, in order to participate in the study, were allowed to have skin-to-skin contact with their babies only once and for at least 15 minutes within the first 4 hours after birth, after the mother and baby had skin-to-skin contact after the baby was born and the baby was breastfed. If the father had any questions about skin-to-skin contact, they were given an explanation, and their questions were answered.
  Interventions: Behavioral: Skin to Skin contact
- Frequent skin-to-skin contact group (FSSC): (Experimental): Fathers in this group, according to the order of participation in the study, were provided skin-to-skin contact with their babies for at least 15 minutes within the first 4 hours after birth, after which skin-to-skin contact was established between the mother and baby after the baby was born and the baby was breastfed and within the first 4 hours after birth. However, skin-to-skin contact with babies by fathers in this group was repeated at least once a day for at least 15 minutes in the hospital until the baby was discharged. After the mother and baby were discharged, fathers were asked to continue skin-to-skin contact at home for at least 15 minutes at least once a day or at least six days a week. In addition, a brochure prepared in accordance with the literature was given to these fathers.
  Interventions: Behavioral: Skin to Skin contact

INTERVENTIONS:
Behavioral: Skin to Skin contact — Fathers are briefed on skin-to-skin: what it is/isn't, why it matters, how to do it, and benefits for father, mother, and baby. Keep the room quiet; close windows to avoid drafts. Do not perform if the father is sleeping. Smokers must not perform while smoking and should do it before smoking when possible. After mother-infant skin-to-skin and breastfeeding, start father-infant contact within four hours of birth. If clothing is unsuitable, provide a surgical gown. Place the diapered infant upright on the father's bare chest. The father supports shoulders and back, maintains eye contact, speaks softly, and touches the baby. Cover both with a blanket; only mother, father, and infant remain, with the researcher silent. Continue at least 15 minutes; end if the father requests care or the infant needs care (diapering, dressing, breastfeeding). Repeat once for the early-contact group and at least daily until discharge for the frequent-contact group; on discharge, remind daily home practice.
  Arms: Early skin-to-skin contact group (ESSC):; Frequent skin-to-skin contact group (FSSC):

SUMMARY:
This randomized, parallel-group clinical trial evaluates whether father-infant skin-to-skin contact improves bonding among healthy term newborns and their fathers in Türkiye. Fathers are randomly assigned to one of three arms that differ in the timing and frequency of skin-to-skin contact (early one-time contact, frequent contact, or standard care). Bonding is assessed with a validated paternal-infant bonding scale at prespecified postpartum time points. The study enrolls fathers of newborns delivered in university and state hospital obstetrics units.

DETAILED DESCRIPTION:
Rationale: Early skin-to-skin contact may facilitate father-infant bonding; experimental evidence in Türkiye is limited.

Design: Interventional, randomized, parallel assignment with three arms:

* Early skin-to-skin contact: a single early skin-to-skin session.
* Frequent skin-to-skin contact: repeated skin-to-skin sessions (e.g., ≥15 minutes per session on most days).
* Standard care: routine postnatal care without a structured skin-to-skin schedule.Participants: Fathers ≥18 years with healthy term singleton newborns.

Assessments: Paternal-Infant bonding is measured using a validated bonding scale at baseline and at a prespecified postpartum time point (e.g., 3 months). Additional baseline questionnaires are collected.

Analysis plan (summary): Group comparisons and exploratory associations will be evaluated per protocol using appropriate statistical tests; full statistical details are provided in the Results section upon completion.

ELIGIBILITY:
Inclusion Criteria:

* Fathers ≥18 years old
* First-time fathers
* At least primary school graduates
* Able to provide ≥15 minutes of skin-to-skin contact within 4 hours of birth
* No communication problems
* Co-resident with their spouses
* Infant: single, healthy newborn at 38-42 weeks' gestation and present with the mother
* (If applicable) Infant birth weight between 2500-4000 g

Exclusion Criteria:

* Fathers who could not be reached during data collection or follow-up
* Separation from the infant for more than one week during follow-up (e.g., hospitalization of the father or infant, long-term work travel)
* Infants requiring special care or with congenital anomalies/serious illness

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2025-02-05 (Actual)

PRIMARY OUTCOMES:
Paternal-Infant Attachment Scale (PIAS) Total Score at 3 Months Postpartum | 3 months postpartum
  Assessed with the Paternal-Infant Attachment Scale (PIAS). The PIAS has 19 items in three subscales and yields a total score from 19 to 95 points; higher scores indicate stronger father-infant bonding. The PIAS is self-reported by fathers at the postpartum assessment.

SECONDARY OUTCOMES:
Patience and Tolerance Subscale Score (PIAS) at 3 Months Postpartum | 3 months postpartum
  Subscale of the PIAS; higher scores indicate stronger bonding. Administered at the postpartum assessment.
Pleasure in Interaction Subscale Score (PIAS) at 3 Months Postpartum | 3 months postpartum
  Subscale of the PIAS; higher scores indicate stronger bonding. Administered at the postpartum assessment.
Affection and Pride Subscale Score (PIAS) at 3 Months Postpartum | 3 months postpartum
  Subscale of the PIAS; higher scores indicate stronger bonding. Administered at the postpartum assessment.
Frequency of Father-Infant Skin-to-Skin Contact (days/week) | Up to 3 months postpartum
  Number of days per week fathers report skin-to-skin contact with their infants, captured by questionnaire at the postpartum assessment.
Daily Minutes of Father-Infant Skin-to-Skin Contact | Up to 3 months postpartum
  Average daily minutes of skin-to-skin contact reported by fathers at the postpartum assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- Çanakkale Onsekiz MArt University Hospital, Çanakkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated and/or analysed during the current study are available on the researcher's computer. The datasets used and/or analysed during the current study are available from the corresponding author upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Derived] Yurdal NEO, Ozsoy S. Effect of skin to skin contact on father infant bonding in a randomized controlled trial. Sci Rep. 2025 Nov 19;15(1):40728. doi: 10.1038/s41598-025-24589-1. PMID 41258333

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-18): https://cdn.clinicaltrials.gov/large-docs/77/NCT07159477/Prot_SAP_000.pdf
  • Informed Consent Form (2023-01-18): https://cdn.clinicaltrials.gov/large-docs/77/NCT07159477/ICF_001.pdf